CLINICAL TRIAL: NCT05414526
Title: Integrating Hypertension and Cardiovascular Diseases Care Into Existing HIV Services Package in Botswana (InterCARE)
Acronym: InterCARE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Botswana (Other)
Responsible Party: Principal Investigator, Mosepele Mosepele, Associate Professor, University of Botswana
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: InterCARE project
Record Dates: First submitted 2022-05-18; First posted 2022-06-10 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: HIV Infections; Hypertension
MeSH Terms: conditions — HIV Infections; Hypertension

STUDY DESIGN:
Intervention Model Description: InterCARE is the name of the package of implementation strategies proposed by the investigators that are intended to integrate cardiovascular care services into existing HIV care systems in Botswana.
  The InterCARE package includes 3 main interventions:
  1. a tailored inter-professional training curriculum on management of CVD risk and HIV
  2. adaptation of the existing electronic health records (PIMS)
  3. adoption of a treatment partner support system.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- InterCARE package (Experimental): The type 2 hybrid effectiveness-implementation study will be cluster randomized trial with 1:1 paired randomization (Intervention arm vs Control arm )Using the coin flip randomization method, one clinic will be randomized to the intervention condition, and one to the control condition.
  Interventions: Other: InterCARE package

INTERVENTIONS:
Other: InterCARE package — The InterCARE package includes:
  1. Healthcare Provider HTN/CVD Curriculum A new HTN curriculum will be developed in collaboration with local stakeholders using KITSO Master trainer program documents (Healthcare provider HIV curriculum), Primary Care Guidelines, HTN/CVD curriculum/protocols trialled in Kweneng District and the CDC Prevention Hypertension Management Curriculum.
  2. Adaptation of HIV care EHR for HTN/CVD care EHR modifications will be done to enhance data collection around HTN/CVD care, with input from MoH.
  3. Patient and treatment partner sessions Clinic staff will provide in-clinic education and counselling on HTN/CVD to all PLWHIV with a diagnosis of hypertension during their routine HIV clinic visit. All patients will be provided a take-home easy-to-read pamphlet on HTN/CVD risk factor management. All PLWHIV will be asked to bring a treatment partner from their social network at the 2nd study visit so that they can practice role-plays with each other.

SUMMARY:
The InterCARE research project proposes to leverage a successful national ART program to develop an effective package to improve the uptake of established effective hypertension and CVD risk factors management interventions among PLWHIV in Botswana and other low- and middle-income countries.

Being the first project of its kind in Botswana, if successful, the InterCARE package could be readily rolled out to health facilities nationwide to diagnose, treat, track, and support the estimated 25-30% Batswana with hypertension.

DETAILED DESCRIPTION:
The InterCARE research project is in 2 phases:

1. Phase 1 is a pilot study to refine the 3 interventions mentioned above. This formative phase will take place between September 2021 and November 2022. Clinics staff will receive training on the management of CVD (and hypertension in particular) in-person or online. Attendees feedback will be sought to improve the curriculum prior to being rolled-out in the next phase of this research project.

   In parallel, the InterCARE Study Team will work with the 2 clinics Information Technology teams to adapt the existing electronic health records with CVD-specific flags, medication lists and laboratory panels.

   Finally, up to 288 participants (PLWHIV) and their treatment partners will be enrolled from those 2 clinics patients lists to pilot the overall InterCARE package.

   The results and experiences from the pilot stage will be assessed and collated to make improvements to each of the 3 intervention in the package. This final set of improved interventions will be the basis of the second phase of the InterCARE research project.

   Phase 1 was successfully completed in November 2022.
2. The InterCARE package will be tested as a cluster randomised trial in 14 clinics around Botswana: 7 clinics will receive the InterCARE package while the remaining 7 clinics will not received any intervention, continuing with the local standard of care, with a target combined recruitment target of 4652 participants overall, to be followed up for 24 months.

Phase 2 is anticipated to take place from January 2023 to July 2025.

ELIGIBILITY:
Inclusion criteria for participants:

* Adults aged 20-75 years old
* Documented HIV-infection on ART
* Confirmed diagnosis of hypertension or elevated blood pressure >140/90mmHg versus >130/80mmHg if they have underlying Diabetes Mellitus or Chronic Kidney Disease
* Receiving regular care at the selected clinics

Exclusion Criteria:

● Positive for HIV-related dementia

Inclusion criteria for participants' treatment partners:

* Adults aged 18 years of age or older
* Selected to be a treatment partner by participant.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4655 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Effectiveness | Every 6 months for 2 years
  Proportion of PLWHIV with diagnosed hypertension receiving anti-hypertensive medication with controlled blood pressure
Implementation | Every 6 months for 2 years
  Proportion of clinic encounters in electronic health records where anti-hypertensive medications are prescribed if indicated, as attained from electronic health records

SECONDARY OUTCOMES:
Reach | Every 6 months for 2 years
  Proportion of PLWHIV who are aware of their hypertension status
Effectiveness | Every 12 months for 2 years
  Decrease in mean systolic blood pressure and mean diastolic blood pressure at 12 and 24 months
Adoption | Every 6 months for 2 years
  Proportion of PLWHIV with hypertension with 10-year cardiovascular risk calculated in the electronic health records
Reach | Every 6 months for 2 years
  Proportion of PLWHIV with diagnosed hypertension receiving anti-hypertensive medication or with BP control not on medications
Maintenance | Every 6 months for 2 years
  Proportion of PLWHIV with HTN enrolled in InterCARE with BP control who maintain blood pressure control in next study visit
Adoption | Every 6 months for 2 years
  Proportion of PLWHIV with HTN enrolled in InterCARE receiving HTN and HIV care in the same clinic visit
Fidelity | Every 6 months for 2 years
  Proportion of PLWH and HTN on medications with correct regimen per national guidelines
Maintenance | Every 12 months for 2 years
  Provider and patient perceptions of ability to maintain a change in blood pressure control:Pre and Post implementation surveys will be used to assess this outcome
Maintenance | At the end of the trial (24 months)
  Proportion of intervention clinics that implemented the three components of InterCARE
Acceptability | At the end of the trial
  Acceptability to patients,mopati and providers (survey and interviews) of the implementation strategy
Effectiveness | Every 6 months for 2 years
  Proportion of PLWHIV with >70% pass on Heart Disease Fact Questionnaire (HDFQ) (health knowledge) .HDFQ score (out of 100):Minimum 0,maximum score 100 :Better Score >70%

CONTACTS AND LOCATIONS:
Overall Officials: Mosepele Mosepele, MD, Principal Investigator — University of Botswana
Locations (3):
- Botswana (3):
  - 14 Infectious Diseases Care centres (IDCCs) nationwide, Gaborone
  - Phitsane-Molopo IDCC Clinic, Pitsane
  - Tonota IDCC Clinic, Tonota

IPD SHARING:
Plan to Share IPD: No
Data recorded as part of the study will be anonymised and will be deposited in a secured archiving facility at the University of Botswana Health Records Unit. Researchers may request access to data as part of transparency and data sharing however this is strictly upon request and will be governed through the required legal office, with at the least, a Data Sharing Agreement in place.
  Further details on this can be found in our Data Management plan.

REFERENCES:
- [Derived] Youssouf N, Mogaetsho GE, Moshomo T, Gaolathe T, Ponatshego P, Ramotsababa M, Molefe-Baikai OJ, Dintwa E, Kiki T, Van Pelt AE, Steger-May K, Bogart LM, Jaffar S, Gala P, Wang D, Seipone K, Bennett K, Hurwitz KW, Kebotsamang K, Hirschhorn LR, Mosepele M. Designing an implementation science clinical trial to integrate hypertension and cardiovascular diseases care into existing HIV services package in Botswana (InterCARE). Trials. 2024 Jul 29;25(1):510. doi: 10.1186/s13063-024-08333-0. PMID 39075506
- [Derived] Moshomo T, Gaolathe T, Ramotsababa M, Molefe-Baikai OJ, Mogaetsho E, Dintwa E, Gala P, Ponatshego P, Bogart LM, Youssouf N, Seipone K, Van Pelt AE, Bennett K, Jaffar S, Ilias M, Tonwe V, Hurwitz KW, Kebotsamang K, Steger-May K, Hirschhorn LR, Mosepele M. Quantitative outcomes of a type 2 single arm hybrid effectiveness implementation pilot study for hypertension-HIV integration in Botswana. Implement Sci Commun. 2024 Jul 22;5(1):80. doi: 10.1186/s43058-024-00620-w. PMID 39039609
- [Derived] Gala P, Ponatshego P, Bogart LM, Youssouf N, Ramotsababa M, Van Pelt AE, Moshomo T, Dintwa E, Seipone K, Ilias M, Tonwe V, Gaolathe T, Hirschhorn LR, Mosepele M. A mixed methods approach identifying facilitators and barriers to guide adaptations to InterCARE strategies: an integrated HIV and hypertension care model in Botswana. Implement Sci Commun. 2024 Jun 20;5(1):67. doi: 10.1186/s43058-024-00603-x. PMID 38902846